CLINICAL TRIAL: NCT05385380
Title: Promoting Safe Motherhood in Ethiopia: A Cluster Randomized Controlled Trial
Brief Title: A Cluster Randomized Controlled Intervention to Improve Institutional Birth Rate in a Rural District of Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Yves Jacquemyn (Other)
Collaborators: Flemish Interuniversity Council (VLIR) (Network); Arba Minch University (Other)
Responsible Party: Sponsor-Investigator, Prof Yves Jacquemyn, Professor, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AMU-IUC-PHD3
Record Dates: First submitted 2022-05-10; First posted 2022-05-23 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Maternal Health Services
Keywords: Antenatal care; Births attended by skilled health providers; Birth Preparedness Plan; Postnatal care

STUDY DESIGN:
Intervention Model Description: A total of 727 pregnant women were recruited and followed up to six months after delivery in this quasi-experimental, two-arm, controlled study. In the intervention group, eligible pregnant women received training to promote safe motherhood, supported by the story "Why Did Mr. X Die, Retold?" and a booklet on working with individuals, families and communities to promote maternal and neonatal health. Pregnant women received counselling (12 sessions/4 sessions per cluster) and biweekly check-ins were performed by community health workers. Pregnant women are encouraged to stay in maternity waiting homes, which have been upgraded to accommodate pregnant women while they wait for their baby to arrive. The control group received standard maternal health information and services as part of the standard health care system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe motherhood Promotion(Educational, Counselling & Training) and maternity waiting homes upgrading (Experimental): 1. Improving the quality of maternal health services in health centers (training for midwives in basic emergency obstetric care and upgrading maternity waiting homes to the level to provide basic accommodation to address access-related barriers
  2. Training community health workers with the aim of improving their knowledge about safe motherhood and about how to prepare a birth plan, including stays in maternity waiting homes
  3. Training pregnant women
  Interventions: Behavioral: Safe motherhood Promotion
- Comparison (No Intervention): The current standard service package

INTERVENTIONS:
Behavioral: Safe motherhood Promotion — Interventions included the training of community members, who subsequently led participatory educational sessions on safe motherhood topics with pregnant females. The project staff identified 2 community health workers and 15 female volunteers from each kebele cluster and trained them as research implementers. The implementers received 2 days of training led by the project team. The project staff and research implementers conducted safe-motherhood training comprising 2 h of information presentations and discussions with pregnant females in the intervention clusters. In addition to the pregnant-female intervention strategy, we also conducted a four-day training programme on clinical skills for local maternal and child healthcare providers in the study area. MWH intervention was also implemented in the intervention group, including upgrades to existing MWH services per national guidelines to standardize services and create a homelike environment for pregnant females.
  Other Names: improving maternity waiting homes
  Arms: Safe motherhood Promotion(Educational, Counselling & Training) and maternity waiting homes upgrading

SUMMARY:
Despite the efforts from the government, maternal healthcare services utilization is far below the recommended level in Ethiopia with a high urban-rural disparity. Currently, two-thirds of pregnant women do not receive the recommended number of antenatal care, more than 50% of births are not attended by skilled birth attendants, and two-thirds of postpartum women do not receive postnatal checks, according to the 2019 EDHS report. There is also evidence that the rate of continuity of maternity care completion is low, implying that pregnant women are not getting the most out of the existing healthcare services. In Ethiopia, the rural communities are scattered over a wide geographic area some with difficult mountains and valleys. Hence, geographic barriers and limited information sources are likely to influence women's access to skilled birth attendance. As part of improving access and overcoming physical or geographical inaccessibility in rural areas, maternity waiting homes; residential lodgings built near healthcare facilities where expectant women near or at term would stay till the onset of labor is one of the measures taken by the Ethiopian government. The majority of the rural populations commonly have a lower perception of health services in general, and many traditional practices support behaviors that are inconsistent with effective health interventions. Thus, there is a challenge concerning behavior (social norms, beliefs, and culture) from the demand side related to utilizing maternity services on top of non/partial functionality of existing waiting homes. Therefore, this research project aimed at promoting access to and utilization of maternal healthcare services utilization in southern Ethiopia.

DETAILED DESCRIPTION:
Health centers and kebeles (villages) in the study setting were randomly assigned to intervention or comparison. We recruited all eligible pregnant women who reside in the respective selected health centres' catchment areas. In the intervention areas, community health workers (unpaid and volunteer women) were identified in consultation with the head of the villages/local leaders/. They received training on safe motherhood, the benefit and importance of maternity homes, identification of local beliefs, traditions and taboos that are barriers to birth preparation, stay in maternity homes and the use of maternal health services. The main functions of these trained community health worker in the intervention clusters include facilitating training sessions for pregnant women, assisting pregnant women in the preparation of birth preparedness plan, supporting pregnant women in starting and sustaining maternity care (prenatal care, skilled delivery and postnatal care). Pregnant women were also trained in the intervention clusters (12 sessions/4 sessions per cluster).

The training of both community health workers and pregnant women was based on a video story titled "Why Did Mr. X Die, Retold?" and a manual on working with individuals, families and communities to improve maternal and neonatal health from the World Health Organization.

After getting permission from the World Health Organization to use the video, we translated it into the local language and used it as an introduction during training. The training was designed based on the findings of preliminary studies and was intended to educate pregnant women about danger signs during pregnancy, labour and the postpartum period, about the birth preparation plan, the benefits and importance of waiting homes. In addition, it also covered how to develop a birth plan that included waiting home with the help of community health workers, as well as correcting misconceptions (belief-related barriers). The intervention was based on principles from the theory of planned behavior and the health belief model. These models were considered to offer direction for what types of variables and processes may be important in shaping maternal health behaviors and thus needed to be addressed in the intervention. The theory of planned behavior is used to explain and predict behavior based on attitudes, norms, and intentions and stipulates that an individual intention to act (behavior) is essentially a function of that individual's attitude toward that behavior and perceptions of social subjective norms. The health belief model which describes how health beliefs interact with modifying factors (e.g., perceived seriousness of problem) to determine health behaviors was also considered in developing the intervention.

The comparison group continued to receive maternal health information and services that are provided as part of the routine healthcare system. Both the baseline and end-line data were managed by trained interviewers using a mobile application supporting Open Data Kit. Data were analyzed through descriptive and inferential statistics (Chi-square test, McNemar tests and multi-level mixed-effects logistic regression analysis). For all analyses, a p-value of <0.05 was considered the level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Those who had resided for at least six months in the selected kebele clusters and had given birth in the five years preceding the survey were included to maintain homogeneity of information exposure. Another criterion for inclusion was a maximum gestational age of 27 weeks (end of second trimester) as participants were required to attend at least two sessions of the proposed promotional intervention before their due date.

Exclusion Criteria:

* Those who met the inclusion criteria but were critically ill at the time of enrolment and/or those who were reluctant to participate were excluded.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The intervention is planned to be delivered to pregnant female.
Enrollment: 727 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
the location of the delivery (home vs. health facility) | through study completion, an average of 9 months
  institutional birth was used to indicate skilled birth attendance as trained health workers do not conduct deliveries outside of health facilities in these areas.
health facility visits after childbirth (postnatal care use) | through study completion, an average of 9 months
  Having visited postnatal clinic after delivery

SECONDARY OUTCOMES:
knowledge of obstetric danger signs | through study completion, an average of 9 months
  Knowledge of birth danger signs was measured using the pregnant females' unprompted responses to the question related to the key danger signs during pregnancy, childbirth and postnatal period
birth preparedness practice | through study completion, an average of 9 months
  Proportion of pregnant women that made prior arrangements for birth and complications

CONTACTS AND LOCATIONS:
Locations (1):
- MEKDES KONDALE Gurara, Arba Minch, Southern Nations Nationalities Regional State, Ethiopia

REFERENCES:
- [Derived] Gurara MK, Draulans V, Jacquemyn Y, Van Geertruyden JP. Evaluation of a community-based intervention package to improve knowledge of obstetric danger signs, birth preparedness, and institutional delivery care utilization in Arba Minch Zuria District, Ethiopia: a cluster-randomized trial. Reprod Health. 2023 Nov 18;20(1):169. doi: 10.1186/s12978-023-01713-w. PMID 37980484